CLINICAL TRIAL: NCT04256018
Title: A Phase 2 Single Center, Single Arm, Open Label Mogamulizumab Combined Upfront With Low Dose Total Skin Electron Beam Therapy (LD TSEBT) in Patients With Mycosis Fungoides (MF) and Sézary Syndrome (SS)
Brief Title: Mogamulizumab + Low-Dose Total Skin Electron Beam Tx in Mycosis Fungoides & Sézary Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-53490; LYMNHL0155 (Other: OnCore); NCI-2020-05893 (Other: NCI Trial Identifier)
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Sezary Syndrome; Mycosis Fungoides
Keywords: CTCL
MeSH Terms: conditions — Sezary Syndrome; Mycosis Fungoides | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LD TSEBT (Experimental): Mogamulizumab with low dose total skin electron beam therapy. •
  LD (12 Gy) TSEBT will be initiated on Cycle 1 Day 2 (± 2 days) of mogamulizumab over 2 to 3 week period per standard of care (SOC), as tolerated. Mogamulizumab (1 mg/kg) will be administered over 60 minutes as follows (per SOC and FDA approved use in MF and SS):
  * Cycle 1 only: Days1; 8; 15; and 22 (± 2 days)
  * Cycle 2 and beyond: Day 1 and Day 15 (± 3 days)
  Interventions: Drug: Mogamulizumab; Radiation: LD TSEBT

INTERVENTIONS:
Drug: Mogamulizumab — Administered 1 mg/kg as an intravenous infusion over at least 60 minutes on Days 1, 8, 15, and 22 of the first 28 day cycle and on Days 1 and 15 of each subsequent cycle.
Radiation: LD TSEBT — Patients will receive total skin dose of 12 Gy fractionated at 4 to 6 Gy per week, for 2-3 weeks
  Other Names: Low-Dose (LD) Total skin electron beam therapy (TSEBT)

SUMMARY:
The purpose of this study is to determine the efficacy of the combination of LD-TSEBT and mogamulizumab in patients with MF and SS. And to evaluate the secondary measures of clinical benefit of the combination therapy and to evaluate the safety and tolerability of the combination in patients with MF and SS.

DETAILED DESCRIPTION:
Primary Objective:To determine the efficacy of the combination of LD TSEBT and mogamulizumab in patients with MF and SS

Secondary Objective: To evaluate the secondary measures of clinical benefit of the combination therapy and to evaluate the safety and tolerability of the combination in patients with MF and SS

ELIGIBILITY:
Inclusion Criteria:

* Stages IB-IV MF or SS

  1. Stages IB-IV MF or SS
  2. At least 1 prior standard-of-care therapy
  3. Prior LD-TSEBT (> 3 months prior) and prior mogamulizumab is allowed, as long as progressive disease (PD) did not occur while on therapy, and did not discontinue due to toxicities
  4. ≥ 18 years of age
  5. ECOG performance status of 0 to 2
  6. All clinically-significant toxic effects of prior cancer therapy resolved to Grade ≤ 1 by the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE, v 5.0).
  7. MF and a known history of non-complicated staphylococcus colonization/infection is eligible provided that stable doses of prophylactic antibiotics continue.
  8. The following minimum wash-out from previous treatments are required (prior to 1st day of treatment), if applicable.

     • ≥ 2weeks for retinoids, interferons, Vorinostat, romidepsin, pralatrexate, or other systemic anti-cancer/CTCL therapies

     • ≥ 2 weeks for phototherapy, local radiation therapy

     • ≥ 2 weeks for topical therapy (including topical steroid, retinoid, nitrogen mustard, or imiquimod)

     • ≥ 12 weeks for total skin electron beam therapy

     • > 12 weeks for alemtuzumab

     • Rapidly progressive malignant disease may be enrolled prior to above periods after discussion with the Protocol Director.
  9. Adequate hematologic function

     • Absolute neutrophil count (ANC) ≥ 1,000 cells/μL (≥ 1,000/mm3)

     • Platelets ≥ 75,000 cells/μL (≥ 75,000/mm3).
  10. Adequate hepatic function

      * Bilirubin ≤ 1.5 times the specific institutional upper limit of normal (ULN). Exception: If Gilbert's syndrome; then ≤ 5 times ULN.
      * Aspartate transaminase (AST) and alanine transaminase (ALT) each ≤ 2.5 x ULN; or ≤ 5.0 x ULN in the presence of known hepatic involvement by CTCL.
  11. Adequate renal function

      • Calculated creatinine clearance ≥ 30 mL/min using the Cockcroft-Gault formula.
  12. If prior allogeneic hematopoietic stem cell transplant (HSCT), then must be free of graft-vs-host disease (GvHD) and receiving immunosuppressive therapy.
  13. Women of childbearing potential (WOCBP) must have a negative pregnancy test.
  14. WOCBP must agree to use effective contraception during the study and for 3 months after the last dose.
  15. Male participants and their female partners of child bearing potential must be willing to use an appropriate method of contraception during the study and for 3 months after the last dose.

      Exclusion Criteria:

  <!-- -->

  1. MF with limited disease (Stage IA) or central nervous system (CNS) disease
  2. Concomitant corticosteroid use. (with the exception that topical steroid and oral prednisone are allowed at ≤ 20 mg/day, if patient has been on a stable dose for at least 2 weeks prior to 1st day of treatment)
  3. Pregnant or breastfeeding
  4. Active autoimmune disease or history deemed by the investigator to be clinically significant
  5. Known human immunodeficiency virus (HIV) positivity; or active hepatitis B or C.
  6. Active herpes simplex or herpes zoster. Those receiving prophylaxis for herpes and who started taking medication at least 30 days prior to the Screening Visit, and have no active signs of active infection, and whose last active infection was more than 6 months ago, may enter the study, and should continue to take the prescribed medication for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 12 months
  Response to treatment will be assessed as the number and proportion of participants who achieve either a complete response (CR) or partial response (PR). The outcome is reported as numbers without dispersion. Clinical response will be assessed as follows.
  * CR: Complete disappearance of all clinical evidence of disease
  * PR: Decrease in size or amount of measurable disease lesions
  * Progressive disease (PD): Worsening of lesions; appearance of new lesions; or recurrence of lesions
  * Stable disease (SD): Disease status that is neither CR, PR, nor PD.

SECONDARY OUTCOMES:
Time-to-Next Significant Treatment (TTNT) | 3 years
  Time-to-next significant treatment (TTNT) will be assessed as the amount of time from starting study treatment through the initiation of any non study systemic therapy. The outcome will be reported as the median TTNT.
Progression free survival (PFS) | 3 years
  Progression free survival (PFS) will be assessed as the amount of time from starting study treatment to progression of disease (PD) or death due to any cause.
Duration of response (DOR) | 3 years
  Duration of response (DOR) will be assessed in those participants who achieve either a complete response (CR) or partial response (PR), and with duration as time to progressive disease or the initiation of a non-study systemic therapy.
  * CR: Complete disappearance of all clinical evidence of disease
  * PR: Decrease in size or amount of measurable disease lesions
  * Progressive disease (PD): Worsening of lesions; appearance of new lesions; or recurrence of lesions
  * Stable disease (SD): Disease status that is neither CR, PR, nor PD.
Patient reported Quality of Life (QoL) | 3 years
  The Skindex 29 survey was used to evaluate the effect of skin conditions on participant's quality of life (QoL). Surveys were administered at the beginning of every treatment cycle and continuing through up to 3 years of treatment. The survey is a 30 item questionnaire with possible answers scored as 1 to 5, with a score of 1 indicating no negative effect, and a score of 5 indicating a constant ("all the time") negative effect. Response ranges are from 30 to 150. The outcome will be reported as the median QoL score with standard deviation.
Treatment-related Adverse Events ≥ Grade 3 | 12 months
  Toxicity will be assessed as adverse events that are severe or greater (≥ Grade 3), and possibly, probably, or definitely related to mogamulizumab or low dose total skin electron beam therapy (LD TSEBT), and occurring within 12 months of starting treatment. The outcome will be reported as the total number of qualifying events, a number without dispersion.
Proportion of Participants With ≥4, ≥6, and ≥12 Months of Response Duration (ORR4, ORR6, and ORR12) | 12 months
  ORR4, ORR6, and ORR12 will be assessed as the proportions of patients who have at least 4, 6, or 12 months of response duration, respectively, among those who achieve either a complete response (CR) or partial response (PR). The outcomes will be reported as numbers without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Kim, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Cancer Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No